CLINICAL TRIAL: NCT00919906
Title: My Scrivener® - Measuring Effectiveness and Dose Response in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Obslap Research LLC (Industry)
Responsible Party: Sue Palsbo, Obslap Research LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 002; #H133S070082
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Asperger's Syndrome; Dyslexia; Cerebral Palsy; Attention Deficit Disorder; ADHD; Traumatic Brain Injury; Stroke
Keywords: haptic; rehabilitation; fine-motor skill; handwriting
MeSH Terms: conditions — Asperger Syndrome; Dyslexia; Cerebral Palsy; Attention Deficit Disorder with Hyperactivity; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handwriting without Tears (No Intervention): Standard practice
- Haptic guidance (Experimental)
  Interventions: Device: My Scrivener(R)

INTERVENTIONS:
Device: My Scrivener(R) — Twenty 20-minute sessions of the Handwriting Without Tears(R) instructional handwriting program, with substitution of hand-over-hand or self-generated repetitive motion writing by computer guided repetitive motion.
  Other Names: My Scrivener; Falcon, by Novint Technologies; Handwriting Without Tears
  Arms: Haptic guidance

SUMMARY:
This study will assess whether a computer haptic peripheral device programmed to provide repetitive motion training is as effective as the same repetitive motion training provided by a human being.

DETAILED DESCRIPTION:
This study builds on a large body of neurological research that uses robot-guided repetitive motion training to induce neuroplasticity and improvements in upper extremity motor skills in adults and children. This research study is looking at handwriting, a fine-motor task that is used daily.

In our study, we want to see if 3-dimensional robotic-assisted repetitive motion training can be a safe and effective intervention for school-age children with fine motor deficits arising from several different impairment origins. Our research construct is: Legible handwriting = function of (tactile feedback, visual feedback, duration, and fine-motor control).

Independent variables:

* Tactile feedback is a continuous variable of force-feedback measured in pounds of force.
* Duration is a continuous variable measured in seconds and number of repetitions.
* Visual feedback is the letter scribed on the paper.

Dependent variable:

* Legible handwriting will be measured by scoring on the Test of Handwriting Skills and the Print Tool™ evaluation.
* Fine motor deficit/control will be measured directly and objectively by quantifying the error between the desired scribing task and the actual scribing task.

The robotic device is an affordable (<$200) computer haptic (the Falcon(R)) that currently is approved by the FCC for home and office. It is *not* approved for medical use. This is an investigational, nonsignificant risk device.

ELIGIBILITY:
Inclusion Criteria:

* Meet the following base prerequisites for writing: orientation to written language; eye-hand coordination, single handed utensil or tool manipulation (BAMF score >= 6), recognize all letters of the alphabet (unless the child has dyslexia).
* Children have illegible printing for their grade, or legible printing but a speed less than the norms for their grade and sex.
* Be able to grasp a pen.
* Be able to speak and understand English.
* Be able to follow instructions.
* Be able to devote at least 20 minutes to the assigned tasks (short breaks will be allowed).
* Be enrolled in school at grade K or above.
* A score lower than 80% on the Print Tool™ or the Cursive Tool.

Exclusion Criteria:

* Unable to pass the informed assent screener.
* Unwilling to sign or mark the informed assent documents.
* Uncontrolled spasticity.
* A BAMF score lower than 6 (includes severe paralysis of the upper extremity).
* Cerebral palsy other than hemiplegia cerebral palsy
* Severe autism or intellectual disabilities that prevent productive interactions with the investigator

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Beery Motor Coordination Subtest | after 20 interventions
Print Tool and Cursive Tool | after 20 interventions
Deviations from desired 3-D writing path | after 5, 10, 15, 20 interventions

SECONDARY OUTCOMES:
Brief Assessment of Fine Motor Skills | after 20 interventions

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Palsbo, PhD, Principal Investigator — Obslap Research LLC
Locations (1):
- Susan Palsbo, Eugene, Oregon, United States

REFERENCES:
- [Background] Bluteau J, Coquillart S, Payan Y, Gentaz E. Haptic guidance improves the visuo-manual tracking of trajectories. PLoS One. 2008 Mar 12;3(3):e1775. doi: 10.1371/journal.pone.0001775. PMID 18335049
- [Background] O'Malley MK, Ro T, Levin HS. Assessing and inducing neuroplasticity with transcranial magnetic stimulation and robotics for motor function. Arch Phys Med Rehabil. 2006 Dec;87(12 Suppl 2):S59-66. doi: 10.1016/j.apmr.2006.08.332. PMID 17140881
- [Background] Volman MJ, van Schendel BM, Jongmans MJ. Handwriting difficulties in primary school children: a search for underlying mechanisms. Am J Occup Ther. 2006 Jul-Aug;60(4):451-60. doi: 10.5014/ajot.60.4.451. PMID 16915876
- [Background] Denton PL, Cope S, Moser C. The effects of sensorimotor-based intervention versus therapeutic practice on improving handwriting performance in 6- to 11-year-old children. Am J Occup Ther. 2006 Jan-Feb;60(1):16-27. doi: 10.5014/ajot.60.1.16. PMID 16541981
- [Background] Palluel-Germain R, Bara F, Hillairet de Boisferon A, Hennion B, Gouagout P, Gentaz E. 2007. A visuo-haptic device - Telemaque - increases kindergarten children's handwriting acquisition. In proceedings of IEEE World Haptics 2007, pp72-77.
- [Background] Marr D, Dimeo SB. Outcomes associated with a summer handwriting course for elementary students. Am J Occup Ther. 2006 Jan-Feb;60(1):10-5. doi: 10.5014/ajot.60.1.10. PMID 16541980
- [Derived] Palsbo SE, Hood-Szivek P. Effect of robotic-assisted three-dimensional repetitive motion to improve hand motor function and control in children with handwriting deficits: a nonrandomized phase 2 device trial. Am J Occup Ther. 2012 Nov-Dec;66(6):682-90. doi: 10.5014/ajot.2012.004556. PMID 23106988
- See also: 3-minute video of the My Scrivener device — http://www.youtube.com/watch?v=niM5gI26U4o